CLINICAL TRIAL: NCT00004178
Title: Phase I Study of T Cells Modified With Chimeric AntiCEA Immunoglobulin-T Cell Receptors (IgTCR) in Adenocarcinoma
Brief Title: Gene Therapy in Treating Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roger Williams Medical Center (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Richard Junghans, Roger Williams Medical Center
Purpose: Treatment
Other Study IDs: CDR0000067388; BIDMC-941101148; NEDH-941101148; NCI-V99-1577
Record Dates: First submitted 2000-01-21; First posted 2004-04-19 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2006-05

CONDITIONS: Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent non-small cell lung cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; stage III cervical cancer; recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; adenocarcinoma of the prostate; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; adenocarcinoma of the stomach; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage III vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; recurrent vaginal cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent endometrial carcinoma; small intestine adenocarcinoma; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage IV non-small cell lung cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; duct cell adenocarcinoma of the pancreas; ovarian undifferentiated adenocarcinoma; adenocarcinoma of the lung; adenocarcinoma of the esophagus; intestinal adenocarcinoma of the stomach; adenocarcinoma of the colon; diffuse adenocarcinoma of the stomach; mixed adenocarcinoma of the stomach; mucinous adenocarcinoma of the colon; signet ring adenocarcinoma of the colon; adenocarcinoma of the rectum; adenocarcinoma of the gallbladder; mucinous adenocarcinoma of the rectum; signet ring adenocarcinoma of the rectum; adenocarcinoma with squamous metaplasia of the gallbladder; adenocarcinoma of the extrahepatic bile duct; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; vaginal adenocarcinoma; vaginal clear cell adenocarcinoma; endometrial adenocarcinoma; cervical adenocarcinoma; adenocarcinoma of the bladder; salivary gland adenocarcinoma; adenocarcinoma of unknown primary; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma; Vaginal Neoplasms; Carcinoma, Hepatocellular; Endometrial Neoplasms; Gallbladder Neoplasms; Bile Duct Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Salivary Gland Neoplasms; Adenocarcinoma of Lung; Adenocarcinoma Of Esophagus

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes

SUMMARY:
RATIONALE: Inserting a gene that has been created in the laboratory into a person's white blood cells may make the body build an immune response to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of gene therapy in treating patients who have cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and maximum tolerated dose of T cells activated in vitro and modified with chimeric anti-CEA immunoglobulin T cell receptors (Ig TCR) in patients with CEA expressing adenocarcinoma.
* Determine the pharmacokinetics of this regimen by the persistence of modified T cells in the blood of these patients.
* Evaluate the immunogenicity of murine sequences in chimeric anti-CEA Ig TCR.
* Assess immunologic parameters which correlate with the efficacy of this regimen in these patients.
* Evaluate, in a preliminary manner, the efficacy of this regimen in patients with CEA bearing tumors.

OUTLINE: This is a dose escalation study.

Peripheral blood lymphocytes (PBL) are harvested. PBL are activated in vitro and then modified with recombinant chimeric anti-CEA immunoglobulin T cell receptors (Ig TCR). Ig TCR modified T cells are reinfused over 30-60 minutes.

The estimated maximum tolerated dose (MTD) is defined as the dose at which 2 of 6 patients experience unacceptable toxicity. If the MTD is not reached within the first cohort, a second cohort of 3 patients then receives 4 doses of modified T cells at a higher dose.

Patients are followed every 2 weeks for 2 months.

PROJECTED ACCRUAL: A total of 6-9 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven CEA expressing adenocarcinoma

  * Serum CEA levels greater than 10 ng/mL
  * Failed standard therapy
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* 0-2

Life expectancy:

* Greater than 2 months

Hematopoietic:

* Not specified

Hepatic:

* No significant hepatic disease
* Bilirubin no greater than 3 mg/dL
* No active clinical disease caused by hepatitis B

Renal:

* No significant renal disease
* Creatinine no greater than 3 mg/dL

Cardiovascular:

* No significant cardiovascular disease

Pulmonary:

* No significant pulmonary disease

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant endocrine, rheumatologic, or allergic disease
* No active clinical disease caused by cytomegalovirus or tuberculosis
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-04; Primary Completion 2000-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard P. Junghans, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States